CLINICAL TRIAL: NCT05958862
Title: Stability of Driving Pressure Changes During "Best Positive End Expiratory Pressure (PEEP)" Trial
Status: Withdrawn | Type: Observational
Why Stopped: Issues with IRB approval. Terminated prior to initiation with no patients enrolled.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Ryan L. Goetz, Pulmonary and Critical Care Medicine Fellow, University of Alabama at Birmingham
Other Study IDs: IRB-300010038
Record Dates: First submitted 2023-06-27; First posted 2023-07-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Acute Respiratory Failure; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to better understand in changes in lung compliance as indicated by driving pressure (a non-invasive marker) following changes in positive end expiratory pressure (PEEP; a standard of care ventilator parameter).

The main question it aims to answer is: The time to stability of driving pressure after a change in PEEP is made Type of study: observational study participant population/health conditions

Participants will undergo a "best PEEP trial" which is a standard intensive care intervention for patients undergoing invasive mechanical ventilation. This involves changing the patient's PEEP and looking for response in driving pressure. This will be done in a more protocolized format and data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >18 years of age
* Undergoing intubation and mechanical ventilation in Medical Intensive Care Unit (MICU) or Medical Critical Care Unit (MCCU) at the University of Alabama Birmingham.

Exclusion Criteria:

* Prisoner
* Pregnant
* Age <18 years of age
* Intensive Care Unit (ICU) team declines participation
* Unstable oxygenation (requiring 100% FiO2 to maintain saturations greater than 90% oxygen saturation following initial PEEP titration by primary team)
* Hemodynamic instability: vasopressor requirement of >0.3 mcg/kg/min of norepinephrine or equivalent
* Pneumomediastinum
* Pneumothorax without chest tube
* Previous enrolled in trial
* Need for immediate travel out of ICU following intubation for procedures, tests

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult medical intensive care patients undergoing invasive mechanical ventilation who meet above inclusion/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Stability of change in Driving Pressure after PEEP manipulation | 10 minutes total
  Our study attempts to find the time point when driving pressure reaches stability. The primary outcome will be the first time point (3 breaths, 30 seconds, 1 minute, 3 minutes, 5 minutes, 10 minutes) where driving pressure is not statistically different from the baseline measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan L Goetz, MD, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: No
No plan to share individual patient level data.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-27): https://cdn.clinicaltrials.gov/large-docs/62/NCT05958862/Prot_SAP_000.pdf